CLINICAL TRIAL: NCT04649060
Title: A Randomized, Controlled, Open-Label Phase 3 Study of Melflufen in Combination With Daratumumab Compared With Daratumumab in Patients With Relapsed or Relapsed-Refractory Multiple Myeloma
Brief Title: Study of Melflufen (Melphalan Flufenamide) in Combination With Daratumumab in Relapsed-Refractory Multiple Myeloma
Acronym: LIGHTHOUSE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study due to financial issues following an FDA request for a partial clinical hold.
Sponsor: Oncopeptides AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OP-108; 2019-002161-36 (EudraCT Number)
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-02

CONDITIONS: Relapsed Multiple Myeloma; Relapsed-Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — melflufen; L-melphalanyl-p-L-fluorophenylalanine ethyl ester; Dexamethasone; daratumumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent Review Committee was planned to be blinded to treatment assignment. Due to the early termination, the response assessments were only done by investigators, not by an independent review committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (melflufen+dexamethasone+daratumumab) (Experimental): Treatment was given in 28-day cycles in an outpatient treatment setting.
  * Melflufen 30 mg intravenous (i.v.) infusion on Day 1 of each cycle
  * Dexamethasone 40 mg per oral (p.o.) weekly (20 mg p.o. weekly if ≥75 years)
  * Daratumumab 1800 mg subcutaneously (s.c.) on Days 1, 8, 15, and 22 in Cycles 1 and 2, on Days 1 and 15 in Cycles 3 to 6, and on Day 1 from Cycle 7
  Interventions: Drug: Melflufen; Drug: Dexamethasone; Drug: Daratumumab
- Arm B (daratumumab) (Active Comparator): Treatment was given in 28-day cycles in an outpatient treatment setting.
  • Daratumumab 1800 mg s.c. on Days 1, 8, 15, and 22 in Cycles 1 and 2, on Days 1 and 15 in Cycles 3 to 6, and on Day 1 from Cycle 7
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Melflufen — Powder for solution for i.v. infusion
  Other Names: Melphalan Flufenamide; Pepaxto; Pepaxti
  Arms: Arm A (melflufen+dexamethasone+daratumumab)
Drug: Dexamethasone — Oral tablets
  Other Names: Dex
  Arms: Arm A (melflufen+dexamethasone+daratumumab)
Drug: Daratumumab — Solution for s.c. injection
  Other Names: Darzalex FASPRO

SUMMARY:
This was a randomized, controlled, open-label, Phase 3 multicenter study which enrolled patients with Relapsed-Refractory Multiple Myeloma (RRMM) who were either double refractory to an Immunomodulatory Drug (IMiD) and a Proteasome Inhibitor (PI) (regardless of the number of prior lines of therapy), or had received at least 3 prior lines of therapy including an IMiD and a PI.

Patients received treatment with melflufen+dexamethasone+daratumumab or daratumumab until documented progressive disease, unacceptable toxicity, or patient/treating physician decision. Patients in the daratumumab treatment arm had the option to receive treatment with melflufen+dexamethasone+daratumumab after confirmed progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* A prior diagnosis of multiple myeloma with documented disease progression after the last line of therapy
* Double refractory to an IMiD and a PI (regardless of the number of prior lines of therapy) or have received at least 3 prior lines of therapy including an IMiD and a PI
* Prior treatment with daratumumab or another anti-CD38 antibody may be allowed under certain circumstances:

  * Achieved at least partial response (PR) and not refractory to an anti-CD38 antibody
  * At least 6 months since the last dose of anti-CD38 antibody
  * Not discontinued anti-CD38 antibody treatment due to related Grade ≥ 3 toxicity
* Male and female of childbearing potential agree to use contraception during the treatment period and at least 3 months after the last dose

Exclusion Criteria:

* Primary refractory disease (i.e., never responded with at least Minimal Response to any prior therapy for multiple myeloma)
* Prior treatment with CD38 CAR-T cell therapy or CD38/CD3 bispecific antibodies
* Any medical condition that may interfere with safety or participation in this study
* Other malignancy diagnosed or requiring treatment within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, carcinoma in-situ of the cervix or breast, or very low and low-risk prostate cancer in active surveillance
* Known or suspected amyloidosis, plasma cell leukemia, or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Known central nervous system (CNS) or meningeal involvement of myeloma
* Prior stem cell transplant (autologous and/or allogenic) within 6 months of initiation of therapy or prior allogeneic stem cell transplantation with active graft-versus-host-disease
* Prior treatment with melflufen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Victorìa Mateos, MD, PhD, Principal Investigator — Complejo Hospitalario de Salamanca
Locations (26):
- Bulgaria (2):
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Clinical Hematology Clinic, Plovdiv
  - Specialized Hospital for Active Treatment of Hematological Diseases, Clinical Hematology Clinic, Sofia
- Czechia (4):
  - University Hospital Brno, Clinic of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Hradec Kralove, 4th Internal Clinic of Hematology, Kralovice
  - University Hospital Ostrava, Clinic of Hematooncology, Ostrava-Poruba
  - General University Hospital in Prague, 1st Internal Clinic - Clinic of Hematology, Prague
- Georgia (2):
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Malkhaz Katsiashvili Multiprofile EMC LTD, Tbilisi
- St. Marien-Hospital Siegen gem. GmbH, Clinic for Hematology, Medical Oncology and Palliative Medicine, Siegen, Germany
- Greece (2):
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - General Hospital of Athens "Evangelismos", Department of Hematology and Lymphoma, Athens
- Oslo University Hospital, Ulleval University Hospital, Oslo Myeloma Center, Oslo, Norway
- Poland (5):
  - Independent Public Healthcare Facility Municipal Hospitals, Teaching Department of Hematology And Prevention of Neoplastic Diseases, Chorzów
  - University Clinical Center, Teaching Department of Hematology and Transplantology, Gdansk
  - Independent Public Healthcare Facility University Hospital in Krakow, Teaching Unit of the Hematology Department, Krakow
  - Nicolaus Copernicus Provincial Multispecialty Oncology and Traumatology Center in Lodz, Lodz
  - St. John of Dukla Oncology Center of Lublin Region, Department of Hematology and Bone Marrow Transplantation, Lublin
- Russia (2):
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - V.D. Seredavin Samara Regional Clinical Hospital, Samara
- Clinical Center of Serbia, Belgrade, Serbia
- Hospital Clinic of Barcelona, Department of Hematology, Barcelona, Spain
- Ukraine (5):
  - Cherkasy Regional Oncology Dispensary, Regional Treatment and Diagnostic Hematology Center, Cherkasy
  - Chernihiv Medical Center of Modern Oncology, Hematology Department, Chernihiv
  - City Clinical Hospital No. 4 City Hematology Center, Dnipro
  - Kyiv City Clinical Hospital No. 9, Hematology Department No. 1, Kyiv
  - National Institute of Cancer, Research Department of Hemoblastosis Chemotherapy and Adjuvant Treatment Methods, Department of Oncohematology with Adjuvant Treatment Methods Group, Kyiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pour L, Szarejko M, Bila J, Schjesvold FH, Spicka I, Maisnar V, Jurczyszyn A, Grudeva-Popova Z, Hajek R, Usenko G, Thuresson M, Norin S, Jarefors S, Bakker NA, Richardson PG, Mateos MV. Efficacy and safety of melflufen plus daratumumab and dexamethasone in relapsed/refractory multiple myeloma: results from the randomized, open-label, phase III LIGHTHOUSE study. Haematologica. 2024 Mar 1;109(3):895-905. doi: 10.3324/haematol.2023.283509. PMID 37646660
- [Derived] Ocio EM, Efebera YA, Hajek R, Straub J, Maisnar V, Eveillard JR, Karlin L, Mateos MV, Oriol A, Ribrag V, Richardson PG, Norin S, Obermuller J, Bakker NA, Pour L. ANCHOR: melflufen plus dexamethasone and daratumumab or bortezomib in relapsed/refractory multiple myeloma: final results of a phase I/IIa study. Haematologica. 2024 Mar 1;109(3):867-876. doi: 10.3324/haematol.2023.283490. PMID 37646657

RESULTS

PARTICIPANT FLOW:
Period: Arm A/Arm B Treatment
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Started | 27 | 27
Treated (There were 6 randomized patients (5 in Arm A and 1 in Arm B) who never received treatment due to failure to meet treatment initiation criteria and/or consent withdrawal.) | 22 | 26
Completed | 0 | 0
Not Completed | 27 | 27
Not completed — Adverse Event | 0 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Progressive Disease | 3 | 12
Not completed — Study Terminated by Sponsor | 17 | 10
Not completed — Patient Request | 1 | 0
Not completed — Failed Criteria for Treatment Initiation | 4 | 1
Not completed — Other | 1 | 0
Period: Crossover (Arm B)
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Started | 0 | 2 (There were 2 patients in Arm B who crossed over and received Melflufen+Dexamethasone+Daratumumab after a confirmed disease progression and received at least one dose of treatment.)
Treated | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab) | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Full Range); unit: years] | 64.5 [43 to 80] | 66.7 [50 to 83] | 65.6 [43 to 83]
Age, Customized [Count of Participants; unit: Participants]
  <65 | 12 | 8 | 20
  65 - ≤75 | 13 | 16 | 29
  >75 | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Full Range); unit: kg] | 79.46 [61.0 to 103.8] | 78.75 [56.3 to 107.6] | 79.1 [56.3 to 107.6]
Height [Mean (Full Range); unit: cm] | 170.4 [151 to 195] | 167.0 [150 to 188] | 168.7 [150 to 195]
Eastern Cooperative Oncology Group (ECOG) score [Count of Participants; unit: Participants] — 0=Normal activity, fully active, able to carry on all pre-disease performance without restriction. 1=Symptoms, but fully ambulatory, restricted in physically strenuous but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    score = 0 | 8 | 6 | 14
    score = 1 | 18 | 15 | 33
    score = 2 | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time from the date of randomization to the date of first documentation of confirmed progressive disease (PD) or death due to any cause, whichever occurred first.
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 27 | 27
months | NA [NA to NA] — The median PFS was not reached in Arm A. There were insufficient numbers of participants with events. | 4.86 [3.38 to NA] — The upper confidence limit was not available due to insufficient numbers of participants with events.
Statistical Analysis 1: Comparison: Arm A (Melflufen+Dexamethasone+Daratumumab) vs Arm B (Daratumumab); Test type: Superiority; p = 0.0032, Log Rank; Hazard Ratio (HR) = 0.184, 95% CI 2-sided [0.052 to 0.650]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Proportion of patients who achieve a best-confirmed response of stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR).
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 27 | 27
percentage of patients | 59.3 [38.8 to 77.6] | 29.6 [13.8 to 50.2]
Statistical Analysis 1: Comparison: Arm A (Melflufen+Dexamethasone+Daratumumab) vs Arm B (Daratumumab); Test type: Superiority; p = 0.03, Cochran-Mantel-Haenszel

3. Secondary Outcome: Duration of Response (DOR)
Description: Time from the first evidence of confirmed assessment of sCR, CR, VGPR or PR to first confirmed disease progression, or death due to any cause. DOR is defined only for patients with a confirmed PR or better.
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 16 | 8
months | NA [NA to NA] — The median DOR was not reached in Arm A and the 95% CI was not available due to insufficient numbers of participants with events. | NA [2.79 to NA] — The median DOR was not reached in Arm B and the upper confidence limit was not available due to insufficient numbers of participants with events.
Statistical Analysis 1: Comparison: Arm A (Melflufen+Dexamethasone+Daratumumab) vs Arm B (Daratumumab); Test type: Superiority; p = 0.525, Log Rank; Hazard Ratio (HR) = 0.418, 95% CI 2-sided [0.026 to 6.693]

4. Secondary Outcome: Best Response
Description: Proportion of patients with sCR, CR, VGPR, PR, Minimal Response (MR), Stable Disease (SD), PD, or non-evaluable (NE).
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 27 | 27
Participants
  Complete Response (CR) | 1 | 0
  Very Good Partial Response (VGPR) | 4 | 3
  Partial Response (PR) | 11 | 5
  Minimal Response (MR) | 3 | 5
  Stable Disease (SD) | 3 | 5
  Progressive Disease (PD) | 1 | 5
  Not Evaluable (NE) | 4 | 4

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The proportion of patients who achieve a best confirmed response of sCR, CR, VGPR, PR, or MR.
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 27 | 27
percentage of patients | 70.4 [49.8 to 86.2] | 48.1 [28.7 to 68.1]
Statistical Analysis 1: Comparison: Arm A (Melflufen+Dexamethasone+Daratumumab) vs Arm B (Daratumumab); Test type: Superiority; p = 0.0997, Cochran-Mantel-Haenszel

6. Secondary Outcome: Duration of Clinical Benefit (DOCB)
Description: Time from first evidence of confirmed assessment of sCR, CR, VGPR, PR, or MR to first confirmed disease progression, or to death due to any cause. DOCB is defined only for patients with a confirmed MR or better.
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 19 | 13
months | NA [NA to NA] — The median DOCB was not reached in Arm A and the 95% CI was not available due to insufficient numbers of participants with events. | NA [3.38 to NA] — The median DOCB was not reached in Arm B and the upper confidence limit was not available due to insufficient numbers of participants with events.
Statistical Analysis 1: Comparison: Arm A (Melflufen+Dexamethasone+Daratumumab) vs Arm B (Daratumumab); Test type: Superiority; p = 0.016, Log Rank; Hazard Ratio (HR) = 0.111, 95% CI 2-sided [0.013 to 0.960]

7. Secondary Outcome: Time to Response (TTR)
Description: Time from randomization to the date of the first documented confirmed response in a patient who has responded with ≥PR.
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 27 | 27
months | 1.8 (1.0) | 1.8 (1.1)

8. Secondary Outcome: Time to Progression (TTP)
Description: Time from randomization to the date of the first documented confirmed PD
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 27 | 27
months | NA [NA to NA] — The median TTP was not reached in Arm A and the 95% CI was not available due to insufficient numbers of participants with events. | NA [4.70 to NA] — The median TTP was not reached in Arm B and the upper confidence limit was not available due to insufficient numbers of participants with events.
Statistical Analysis 1: Comparison: Arm A (Melflufen+Dexamethasone+Daratumumab) vs Arm B (Daratumumab); Test type: Superiority; p = 0.0187, Log Rank; Hazard Ratio (HR) = 0.231, 95% CI 2-sided [0.063 to 0.846]

9. Secondary Outcome: Time to Next Treatment (TTNT)
Description: Time from randomization to the date of next anti-myeloma treatment or until death.
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 27 | 27
months | 11.04 [NA to NA] — The 95% CI was not available due to insufficient numbers of participants with events. | NA [4.40 to NA] — The median TTNT was not reached in Arm B and the upper confidence limit was not available due to insufficient numbers of participants with events.
Statistical Analysis 1: Comparison: Arm A (Melflufen+Dexamethasone+Daratumumab) vs Arm B (Daratumumab); Test type: Superiority; p = 0.0384, Log Rank; Hazard Ratio (HR) = 0.224, 95% CI 2-sided [0.047 to 1.056]

10. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to death due to any cause.
Time Frame: From the date of randomization until the end of study (approximately 12 months).
Population: Analysis was performed using the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab)
Number analyzed (Participants) | 27 | 27
months | 11.04 [NA to NA] — The 95% CI is not available due to insufficient numbers of participants with events. | NA [NA to NA] — The median OS was not reached in Arm B and the 95% CI was not available due to insufficient numbers of participants with events.
Statistical Analysis 1: Comparison: Arm A (Melflufen+Dexamethasone+Daratumumab) vs Arm B (Daratumumab); Test type: Superiority; p = 0.3721, Log Rank; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.086 to 2.569]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the start of study treatment until 30 days after the last dose of study drug or initiation of subsequent therapy whichever occurred first. Serious AEs (SAEs) were collected from signing of the informed consent form (ICF) until 30 days after the last dose of study treatment or initiation of subsequent therapy whichever occurred first. The maximum duration of treatment was 48 weeks, and the maximum duration of AEs/SAEs collection was 48 weeks + 30 days.
Description: AE definition: An AE is any untoward medical occurrence in a patient or clinical study patient, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
  AEs are grouped by MedDRA system organ class (SOC) and preferred term (PT).
Groups:
- Crossover (From Arm B to the Same Treatment as Arm A): Patients in Arm B were allowed to crossover and receive the same treatment as Arm A after a confirmed disease progression (2 patients crossed over).
Arm/Group | Arm A (Melflufen+Dexamethasone+Daratumumab) | Arm B (Daratumumab) | Crossover (From Arm B to the Same Treatment as Arm A)
All-Cause Mortality (participants affected / at risk) | 2/22 | 3/26 | 1/2
Serious Adverse Events (participants affected / at risk) | 6/22 | 12/26 | 1/2
Other Adverse Events (participants affected / at risk) | 21/22 | 22/26 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Melflufen+Dexamethasone+Daratumumab) (N=22) | Arm B (Daratumumab) (N=26) | Crossover (From Arm B to the Same Treatment as Arm A) (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Melflufen+Dexamethasone+Daratumumab) (N=22) | Arm B (Daratumumab) (N=26) | Crossover (From Arm B to the Same Treatment as Arm A) (N=2)
Pneumonia (Infections and infestations) | 2 | 3 | 1
Infection (Infections and infestations) | 2 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 13 | 8 | 1
Anaemia (Blood and lymphatic system disorders) | 12 | 7 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 4 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 0
Fatigue (General disorders) | 2 | 0 | 0
Neutrophil count decrease (Investigations) | 3 | 0 | 0
Platelet count decrease (Investigations) | 2 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was put on clinical hold and later discontinued prematurely. Due to this, there is limited data available, and data cleaning was not done according to the original plan. Due to the early termination, the response assessments were done by investigators, not by an independent review committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT04649060/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT04649060/SAP_001.pdf